CLINICAL TRIAL: NCT05341934
Title: Evaluative Conditioning: A Brief Cognitive Intervention Aimed to Modify Addiction Behaviour of Alcohol-dependent Patients
Acronym: CEAlcool
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Inclusion/ Study never begin
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A02120-53
Record Dates: First submitted 2020-07-15; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Intervention to Modify Addiction Behaviour of Alcohol-dependent Patients
Keywords: evaluative conditionning, addiction, alcohol, patients
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conditionning (Active Comparator)
  Interventions: Other: Evaluative Conditionning Task
- Placebo (Placebo Comparator)
  Interventions: Other: Evaluative Conditionning Task

INTERVENTIONS:
Other: Evaluative Conditionning Task — A word will appear in one of the four quadrants on the computer screen. They will have to answer the word as quickly as possible by pressing the space bar. They will also be told that an image will be displayed briefly (400 ms) in the same quadrant by pressing the answer key. This procedure will be repeated for 120 trials: 30 trials with alcohol-related Conditional Stimulus (CS), 30 trials with CS related to non-alcoholic beverages and 60 trials with the CS of filling. The CS referring to alcohol will be the words Beer, Wine …; The CS referring to soft drinks will be the words Coca-Cola, Fanta… and Filling CS referring to vegetables and fruits will be: Apple, Banana…In experimental conditions, alcohol-related CS will be followed by negative Unconditional Stimuli (US) (images from the International Affective Picture System (Lang, Bradley, & Cuthbert, 1997)), CS referring to soft drinks linked to positive images and CS referring to fruits and vegetables will be linked to neutral US.
  Other Names: Implicit Association Task; Subliminal Attitude Misattribution Procedure

SUMMARY:
Evaluative Conditioning: A Brief Cognitive Intervention Aimed to Modify Addiction Behaviour of Alcohol-dependent Patients

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study will be patients:
* With an alcohol use disorder according to DSM 5
* Follow-up at the Laborit Hospital Center
* Aged between 18 and 70 years with informed consent after receiving written information
* Engaged in a process to reduce alcohol consumption
* With a score of MOCA> 20
* Whose mother tongue is French
* Patients benefiting from social security or benefiting from it through a third party in accordance with the french law on research involving the human person.

Exclusion Criteria:

* - Patient with less than 6 Heavy Drinking Days in the month
* Patient with Schizophrenia
* Patient with bipolar disorder Type 1
* Patient with Korsakoff syndrome or degenerative neurological disorder
* Patient with hearing impairment, uncorrected visual impairment
* Patient under curatorship or guardianship
* Patient with addiction to another substance other than tobacco
* Patient already enrolled in another interventional study
* Pregnant or nursing woman
* Patient with difficulties of expression or comprehension in French
* Patients in emergency situations or unable to give their consent.

Output Criteria:

* Patient who has manifested verbally or in writing, the desire to leave the study in progress.
* Patient who will be hospitalized during the study for a problem related to his addiction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The reduction of automatic or implicit associations of Alcohol with positive affect. | baseline
  It will be evaluated by calculating the difference between the scores of the IAT task before and after the Evaluative Conditioning.

SECONDARY OUTCOMES:
The reduction in the total amount of alcohol consumed | week 2
  The reduction in the total amount of alcohol consumed (TAC: Total Alcohol Consumption) as well as the number of Heavy Drinking Day (HDD) over the 12-week period following treatment, with respect to the baseline time.
  The baseline time is the week before randomization. Consumption of alcohol (total quantity and consumption habits) during this period will be considered as a baseline.
  The HDD corresponds to the days of consumption of more than 60 grams of pure alcohol (men) or 40 grams (women).
The reduction in the total amount of alcohol consumed | month 3
  The reduction in the total amount of alcohol consumed (TAC: Total Alcohol Consumption) as well as the number of Heavy Drinking Day (HDD) over the 12-week period following treatment, with respect to the baseline time.
  The baseline time is the week before randomization. Consumption of alcohol (total quantity and consumption habits) during this period will be considered as a baseline.
  The HDD corresponds to the days of consumption of more than 60 grams of pure alcohol (men) or 40 grams (women).

CONTACTS AND LOCATIONS:
Overall Officials: JAAFARI NEMATOLLAH, PROFESSOR, Principal Investigator — Centre Hospitalier Henri Laborit
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided